CLINICAL TRIAL: NCT03523091
Title: Is Less More? Does Decreasing OnabotulinumtoxinA Injection Sites in the Bladder Increase Patient Satisfaction While Maintaining Efficacy?
Brief Title: OnabotulinumtoxinA Bladder Injection Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Larry Sirls, Attending Urologist, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-119
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome; Urinary Urgency; Urinary Incontinence; Urinary Frequency/Urgency; Urinary Bladder, Overactive
Keywords: OnabotulinumtoxinA; Bladder Injections
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: 2 arm parallel study with 1 to 1 randomization
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 3 Injection Sites (Experimental): OnabotulinumtoxinA 100Unit injection into 3 sites throughout the bladder
  Interventions: Drug: OnabotulinumtoxinA 100Unit Injection
- 10 Injection Sites (Experimental): OnabotulinumtoxinA 100Unit injection into 10 sites throughout the bladder
  Interventions: Drug: OnabotulinumtoxinA 100Unit Injection

INTERVENTIONS:
Drug: OnabotulinumtoxinA 100Unit Injection — Initial treatment with the option of repeat injections every 3 months
  Other Names: Botox

SUMMARY:
Patients with overactive bladder (OAB) will be randomly assigned (like a flip of a coin) to receive 100 units of onabotulinumtoxinA injected into the bladder at either 3 sites or 10 sites. Patient satisfaction and the effectiveness of the medication will be evaluated.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a common condition which often has a negative impact on health related quality of life. Primary and secondary treatments include behavior modification, pelvic floor physical therapy, and OAB medications. OnabotulinumtoxinA (BTX) is a well-established third line therapy for refractory OAB.

BTX has transitioned over the years from a procedure conducted in the operating room to one that is commonly done in the clinic or physician office. While ten injection sites is commonly practiced, there has been continuing interest in reducing the number of injection sites to make the technique more tolerable and more efficient.

In this study, refractory OAB patients will be randomized to receive 100 units of BTX over 3 or 10 injection sites. The investigators hypothesize that decreasing the number of injection sites may improve patient tolerability and satisfaction with this office-based procedure and potentially reduce the rates of adverse events including hematuria and urinary tract infection.

ELIGIBILITY:
Inclusion Criteria:

* Women and men, 18 years of age or older
* Self-reported failed conservative care of behavioral modifications and/or oral medications for the treatment of OAB
* Average urinary frequency of > 8 voids per day as recorded on initial 3-day voiding diary
* Self-reported bladder symptoms > 3 months
* Discontinued antimuscarinics/beta-3 agonists for > 2 weeks prior to study enrollment. May restart antimuscarinics/beta-3 agonists if indicated > 6 weeks after Botox injections.
* Capable of giving informed consent
* Capable and willing to follow all study-related procedures
* Previous OnabotulinumtoxinA injection at least three months prior to study enrollment.

Exclusion Criteria:

* Pregnant or planning to become pregnant during study duration
* Diagnosis of neurogenic bladder with the exception of highly functioning stroke patients
* If a patient has had a previous neuromodulation device placed, it will have to be turned off for 2 weeks for a washout period and remain off throughout the study
* Previous non-responders to onabotulinumtoxinA (BTX) therapy
* Patient cannot be receiving percutaneous nerve stimulation (PTNS) therapy. If patient is receiving PTNS, they need to stop for 1 month prior to entering the study.
* Refusal to self-catheterize or have indwelling catheter in the event of urinary retention
* Use of investigational drug/device therapy within past 4 weeks
* Participation in any clinical investigation involving or impacting gynecologic, urinary or renal function within past 4 weeks
* Current or past history of any physical condition that, in the investigator's opinion, might put the subject at risk or interfere with study results interpretation
* Pelvic radiation treatment
* Known hypersensitivity to OnabotulinumtoxinA.
* Previous infection at OnabotulinumtoxinA injection site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Sirls, MD, Principal Investigator — Beaumont Hospital-Royal Oak
Locations (1):
- Beaumont Hospital-Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will not be available

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3 Injection Sites | 10 Injection Sites
Started | 1 | 5
Completed | 0 | 1
Not Completed | 1 | 4
Not completed — Lower dose due to elevated post void residual (PVR) | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Increase Botox dose | 0 | 1

BASELINE CHARACTERISTICS:
Population: Of the initial 6 subjects consented, 1 subject was randomized to the 3 injection site arm and 5 were randomized to the 10 injection site arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 Injection Sites | 10 Injection Sites | Total
Number analyzed (Participants) | 1 | 5 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 3
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 5 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 4 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 5 | 6
Baseline number of voids [Mean (Standard Deviation); unit: Voids] — Participants will be asked to complete a 3-day voiding diary. On the diary participants will record the number of occurrences of incontinence episodes over a 24 hour period for 3 consecutive days.
  Voids | 14 (0) | 14.9 (6.02) | 14.8 (5.4)
Baseline number of urge incontinence episodes [Mean (Standard Deviation); unit: Urge incontinence episodes] — Participants will be asked to complete a 3-day voiding diary. On the diary participants will record the number of urge incontinence episodes over a 24 hour period for 3 consecutive days.
  Urge incontinence episodes | 21 (0) | 20.6 (12.1) | 20.7 (10.8)
Baseline number of stress incontinence episodes [Mean (Standard Deviation); unit: Stress incontinence episodes] — Participants will be asked to complete a 3-day voiding diary. On the diary participants will record the number of stress incontinence episodes over a 24 hour period for 3 consecutive days
  Stress incontinence episodes | 0 (0) | 0.2 (0.4) | 0.17 (0.4)
Baseline Symptom Bother [Mean (Standard Deviation); unit: score on a scale] — Per the Overactive Bladder Questionnaire-Short Form (OABq-SF). This validated measure evaluates overactive bladder symptom severity and health related quality of life. For each question, participants will answer how bothered they are by their urinary symptoms from "not at all" (1), "a little bit" (2), "somewhat" (3), "quite a bit" (4), "a great deal" (5), and "a very great deal" (5). Each question will be scored. Scores range from 19-114. The higher the score the greater perceived degree of bladder symptom bother.
  score on a scale | 64 (0) | 87.4 (14.7) | 83.5 (16.2)
Baseline severity of urine leakage [Mean (Standard Deviation); unit: score on a scale] — Per the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF). This validated questionnaire provides a measure to assess the impact of symptoms of incontinence on quality of life and outcome of treatment. Question items include frequency of urinary incontinence, amount of leakage, overall impact of urinary incontinence, and a self-diagnostic item. Scoring is between 0-21 with greater values indicating increased severity.
  score on a scale | 16 (0) | 15 (8.5) | 15.2 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Incontinence Episodes Per Day
Description: Participants will be asked to complete a 3-day voiding diary. On the diary participants will record the number of occurrences of voids over a 24 hour period for 3 consecutive days. Number of voids at 3 months are recorded.
Time Frame: 3 months after the initial injection
Population: Due to the small number of participants statistical analysis was limited. 3 participants completed 3 month diary data.
Measure: Mean (Standard Deviation); unit: Incontinency episodes
Arm/Group | 3 Injection Sites | 10 Injection Sites
Number analyzed (Participants) | 1 | 2
Incontinency episodes | 0 (0) | 15.5 (21.9)

2. Secondary Outcome: Degree of Bladder Symptom Bother
Description: Per the Overactive Bladder Questionnaire-Short Form (OABq-SF). This validated measure evaluates overactive bladder symptom severity and health related quality of life. For each question, participants will answer how bothered they are by their urinary symptoms from "not at all" (1), "a little bit" (2), "somewhat" (3), "quite a bit" (4), "a great deal" (5), and "a very great deal" (5). Each question will be scored. Scores range from 19-114. The higher the score the greater perceived degree of bladder symptom bother.
Time Frame: 3 months after the initial injection
Population: Due to the small number of participants data analysis was limited. 3 participants completed data at 3 months.
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | 3 Injection Sites | 10 Injection Sites
Number analyzed (Participants) | 1 | 2
score on scale | 23 (0) | 43 (26.9)

3. Secondary Outcome: Severity of Urine Leakage
Description: Per the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF). This validated questionnaire provides a measure to assess the impact of symptoms of incontinence on quality of life and outcome of treatment. Question items include frequency of urinary incontinence, amount of leakage, overall impact of urinary incontinence, and a self-diagnostic item. Scoring is between 0-21 with greater values indicating increased severity.
Time Frame: 3 months after the initial injection
Population: Due to small number of participants data analysis was limited. 3 participants had data at 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 Injection Sites | 10 Injection Sites
Number analyzed (Participants) | 1 | 2
score on a scale | 3 (0) | 7.5 (7.5)

4. Secondary Outcome: Change in Overactive Bladder Symptoms
Description: Per the Global Response Assessment (GRA). Participants will assess overall how their OAB symptoms/condition changed since starting the study. Participants will select, "Markedly worse" (1), "Moderately worse" (2), "Mildly worse" (3), "Same (unchanged)" (4), "Slightly improved" (5), "Moderately improved" (6), or "Markedly improved" (7). Scores are from 1-7 with a greater score indicating a greater improvement of symptoms. Numbers of participants reporting each assessment will be reported.
Time Frame: 3 months after the initial injection
Population: Due to a small number of participants data analysis was limited. 3 participants completed GRA data at 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Injection Sites | 10 Injection Sites
Number analyzed (Participants) | 1 | 2
Participants
  Markedly Improved | 1 | 0
  Moderately Improved | 0 | 0
  Slightly Improved | 0 | 1
  No change | 0 | 0
  Slightly Worse | 0 | 1
  Moderately Worse | 0 | 0
  Markedly Worse | 0 | 0

5. Secondary Outcome: Overall Patient Pain Tolerability With Treatment
Description: Per the Visual Analog Scale (VAS). Participants will record the amount of pain of performing the treatment on a Visual Analog Scale from 0 (no pain) to 10 (worst pain imaginable). Visual analog scores will be gathered at the end of the injection visit.
Time Frame: After the initial injection
Population: 6 subjects completed baseline VAS scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3 Injection Sites | 10 Injection Sites
Number analyzed (Participants) | 1 | 5
score on a scale | 2 (0) | 3 (1.10)

6. Secondary Outcome: Overall Voiding Symptoms at 3 Months
Description: Per the 3-day voiding diary. Participants will be asked to complete a 3-day voiding diary. On the diary participants will record the number of occurrences of voids, urge and stress incontinence episodes over a 24 hour period for 3 consecutive days.
Time Frame: 3 months after the initial injection
Population: Due to small number of participants data analysis was limited. 3 subjects had data available for 3 month timepoints.
Measure: Mean (Standard Error); unit: Episodes
Arm/Group | 3 Injection Sites | 10 Injection Sites
Number analyzed (Participants) | 1 | 2
Episodes
  Average number of voids | 12.6 (0) | 13.2 (2.6)
  Urge incontinence episodes | 0 (0) | 11 (15.6)
  Stress incontinence episodes | 0 (0) | 1.5 (2.1)

7. Secondary Outcome: Safety of Bladder Injections
Description: Frequency and severity of study-related adverse events
Time Frame: At study completion, 3 months after the initial injection
Population: 3 participants completed the study through the 3 month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Injection Sites | 10 Injection Sites
Number analyzed (Participants) | 1 | 2
Participants
  Post-void residual over 300 ml, severity mild | 1 | 0
  Urinary tract infection, severity mild | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through study completion, the last study visit was at 3 months.
Arm/Group | 3 Injection Sites | 10 Injection Sites
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/5
Other Adverse Events (participants affected / at risk) | 1/1 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 Injection Sites (N=1) | 10 Injection Sites (N=5)
Post-void resisdual over 300 cc (300 mL) (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT03523091/Prot_SAP_002.pdf
  • Informed Consent Form (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT03523091/ICF_001.pdf